CLINICAL TRIAL: NCT04960956
Title: Glycosylation of Exosomes in Prostate and Urothelial Carcinoma
Status: Terminated | Type: Observational
Why Stopped: Could not identify a replacement Principal Investigator.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Roberto Pili, Associate Dean for Cancer Research and Integrative Oncology, University at Buffalo
Other Study IDs: IUSCC-0588
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer; Urothelial Carcinoma
Keywords: Glycosylation; Urinary Exosomes; Exosome-derived Glycans
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample collection, handling, and storage requirements
  * Collect at least 40-50 mL of fresh fasting urine (Note: up to 200 mL from each subject can be used for this study)
  * Within two hours of collection, add one tablet containing protease inhibitor cocktail and 0.5 mL of 2% sodium azide solution (weight to volume in water) to the sample for preventing bacterial growth (both additives provided by the Novotny Glycoscience Laboratory). Close the cap and mix gently by hand until the additives have dispersed into the urine sample.
  * Label the sample with the study ID, subject ID, date and time of collection
  * Store at -80°C
  * Batch-ship samples on dry ice to:
  Professor Milos Novotny IU Department of Chemistry 800 E. Kirkwood Ave. Bloomington, IN 47405 Phone: 812-855-4532
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect a urine sample from patients with prostate and urothelial (bladder) cancer and healthy volunteers who do not have cancer, so that researchers can perform studies on microcellular structures called exosomes that may eventually lead to a new type of urinary biomarker test for prostate and urothelial cancer.

DETAILED DESCRIPTION:
This is a one-time participation, banking study of up to 40 subjects (10 prostate, 10 urothelial, 20 without cancer). Subjects must meet eligibility at the time of informed consent and will donate approx. 200mL of urine sample.

Primary Objective:

To develop alternative and efficient urinary exosome isolation and glycan analysis approaches for especially large glycan structures, including their isomers present at low levels, which will particularly enhance current analytical technology.

To provide further testing of the current microfluidic-based approaches developed to screen glycan samples which this additional specimen will provide to assess whether the current analytical techniques are robust enough to handle this type of sample with sufficient resolution and sensitivity for useful analytical information.

To compare alterations in exosome-derived glycans in adults with prostate and urothelial carcinoma in comparison with the exosome-derived glycans in age-matched healthy adults for assessment of findings to explore if the tools could be applied for future study toward a liquid biopsy test.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Willingness to donate a fasting urine sample for research Patient Cohort

   1. Histologically confirmed prostate or urothelial carcinoma
   2. Localized disease
   3. No neoadjuvant chemotherapy for disease Healthy Volunteer Cohort

   <!-- -->

   1. Healthy volunteers must not have prostate or urothelial carcinoma

Exclusion Criteria:

1. Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males ≥ 18 years old at the time of informed consent
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
The concentration of urine spermine in the diagnosis of prostate and urothelial cancer | Baseline (one-time point)
  xFresh urine will be collected for MALDI-TOF analysis to detect the concentration of exosome-derived glycans in the urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided